CLINICAL TRIAL: NCT07141615
Title: Clinical Observation of Qingwei Huazhuo Decoction (Product: Jinsaiyu) in Improving Children With Precocious Puberty of Phlegm-Dampness Internal Accumulation Type
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Sunwen, Chief Physician, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FDCH-ZY-2025162
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Precocious Puberty
Keywords: precocious puberty; Qingwei Huazhuo Decoction
MeSH Terms: conditions — Puberty, Precocious | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group is administered Qingwei Huazhuo Decoction therapy and diet and exercise education for a period of six months.
  Interventions: Combination Product: Qingwei Huazhuo Decoction: Mulberry leaf powder, lotus leaf powder, malt powder, hawthorn powder, Poria cocos powder, gardenia powder, dried tangerine peel powder, licorice powder, momordica grosvenor; Behavioral: diet and exercise education
- Control group (Experimental): diet and exercise education
  Interventions: Behavioral: diet and exercise education

INTERVENTIONS:
Combination Product: Qingwei Huazhuo Decoction: Mulberry leaf powder, lotus leaf powder, malt powder, hawthorn powder, Poria cocos powder, gardenia powder, dried tangerine peel powder, licorice powder, momordica grosvenor — On the basis of receiving dietary and exercise education, the pediatric patients were given the Qingwei Huazhuo Decoction orally.
  Composition:Mulberry Leaf Powder, Lotus Leaf Powder, Germinated Barley Powder, Hawthorn Powder, Poria Mushroom Powder, Cape Jasmine Fruit Powder, Tangerine Peel Powder, Licorice Root Powder, Monk Fruit Powder.
  Administration Method:Take one sachet each time, add 150ml of warm boiled water, stir well, and drink.
  Treatment Course:The first-stage course lasts for 12 weeks.For participants in the experimental group who have completed the first 12-week stage, they may continue to take the Qingwei Huazhuo Decoction orally for another 12 weeks
  Arms: Intervention group
Behavioral: diet and exercise education — ① Dietary Education With reference to the Balanced Diet Pagoda for School-Age Children Aged 6-10 Years in the Chinese Dietary Guidelines for School-Age Children (2022), the children were required to record their daily diet and complete a dietary diary.
  ② Exercise Education
  Children were advised to accumulate at least 60 minutes of moderate-to-vigorous physical activity (MVPA) daily, mainly consisting of aerobic exercise. The specific requirements were as follows:
  1.3-5 sessions of aerobic exercise per week; 2.2-3 sessions of resistance exercise per week; 3.Daily screen time limited to less than 2 hours. The parents were asked to record their children's daily completion of the above requirements.

SUMMARY:
Clinical Observation of Qingwei Huazhuo Decoction (Product: Jinsaiyu) in Improving Children With Precocious Puberty of Phlegm-Dampness Internal Accumulation Type

ELIGIBILITY:
Inclusion Criteria:

* 1. With reference to the diagnostic criteria for incomplete precocious puberty (isolated premature thelarche) in *Expert Consensus on the Diagnosis and Treatment of Central Precocious Puberty (2022)* and *Modern Pediatrics Diagnosis and Treatment*, the following requirements must be met: (1) Female children with initial symptoms of unilateral or bilateral breast development, without other signs of sexual development; (2) No accelerated growth and bone age not exceeding the actual age by 1 year; (3) No vaginal bleeding; (4) Plasma estradiol (E2) and follicle-stimulating hormone (FSH) levels within the reference range or slightly elevated.
* 2. Based on the doctor's clinical judgment, the traditional Chinese medicine (TCM) syndrome type conforms to the diagnostic criteria for phlegm-dampness internal accumulation syndrome. With reference to the syndrome classification criteria in *Guidelines for Integrated Traditional Chinese and Western Medicine Diagnosis and Treatment of Pediatric Precocious Puberty (2023 Edition)*, the diagnosis can be made if the child meets 2-3 or more symptoms of any syndrome type, and the tongue and pulse conditions are basically consistent with the syndrome. Details of the syndrome are as follows: Phlegm-dampness internal accumulation: The child has premature appearance of secondary sexual characteristics, which may be accompanied by excessive consumption of fatty and sweet foods, obesity, heavy sensation in limbs, being quiet and inactive, sticky sensation in the mouth, red tongue with thick and greasy coating, and slippery and rapid pulse.
* 3. Obtain the informed consent form signed by the legal guardian of the subject.

Exclusion Criteria:

* 1. Children with peripheral precocious puberty or central precocious puberty (idiopathic and secondary);
* 2. Children with other severe underlying diseases, including but not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidneys, liver, gastrointestinal tract, respiratory system, metabolic system, and skeletal system;
* 3. Those allergic to any component of Qingwei Huazhuo Recipe (Product: Jinsaiyu);
* 4. Those currently participating in other clinical trials or who have participated in other clinical trials within the past 3 months;
* 5. Children judged by researchers to have poor compliance and are not suitable for entering this study.

Ages: 5 Years to 8 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 94 (Estimated)
Dates: Start 2025-09-22 (Estimated); Primary Completion 2027-11-16 (Estimated); Study Completion 2027-12-16 (Estimated)

PRIMARY OUTCOMES:
breast nucleus diameter | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Measured by the attending physician using a straightedge

SECONDARY OUTCOMES:
Bone age | The measurement times are before the start of the experiment and the 24th week after the start.
  Bone age is determined by radiologists in our hospital who take a posteroanterior radiograph of the left hand and judge the bone age according to the Greulich-Pyle (GP) atlas method.
Traditional Chinese Medicine syndrome score | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Based on the *Guidelines for Integrated Traditional Chinese and Western Medicine Diagnosis and Treatment of Pediatric Precocious Puberty (2023 Edition)* and clinical experience, the Traditional Chinese Medicine (TCM) syndrome scores were screened and determined.

OTHER OUTCOMES:
Testosterone | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Testosterone(nmol/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
PRL | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Prolactin(mIU/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
Estradiol | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Estradiol(pmol/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
FSH | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Follicle-Stimulating Hormone(U/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
LH | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Luteinizing Hormone(U/L, detected from the blood) Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.
Height | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  The height is measured and obtained by the physician. Place the mechanical height measuring device horizontally on a flat surface, against a wall, and calibrate the height measuring device reading. Instruct the examinee to stand barefoot on the base plate of the height measuring device, facing away from the pillar. When the doctor moves the height measuring device, he holds the handle of the height measuring device, moves horizontally, tries to keep the head upright, and keeps the body and limbs naturally straight. For hair knots and braids that are not convenient to measure height, they should be untied and headwear should be removed. The horizontal pressure plate should be in contact with the head, and the tightness should be moderate. The data is read in cm units and is accurate to 0.1.
Weight | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  The weight is measured and obtained by the physician. Place the electronic scale flat on the ground, calibrate the scale reading, instruct the examinee to empty their bowels and bladder, wear light clothing and stand barefoot naturally in the center of the electronic scale pedal, keep the body stable, record the data, the unit is kg, and the value is accurate to 0.1.
Waist-Hip Ratio | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Use a flexible, non-elastic anthropometric tape (mm-scale) and have the subject stand upright (feet shoulder-width apart, arms relaxed, abdomen relaxed) in lightweight, form-fitting clothing.
  For waist circumference: Mark the midpoint between the costal arch's inferior margin and iliac crest's superior border (umbilicus as alternative if unclear). Wrap the tape horizontally here-level, skin-adherent, no subcutaneous compression. Record to 0.1 cm at end of normal expiration; average 2-3 readings.
  For hip circumference: Locate the gluteal region's widest transverse diameter (confirmed posteriorly/laterally). Wrap tape horizontally here (level, flat). Record to 0.1 cm; average 2-3 readings.
  Compute WHR as mean waist ÷ mean hip (decimal, e.g., 85.2 cm ÷ 102.5 cm ≈ 0.83). Trained personnel must conduct measurements to reduce inter-observer variation.
Uterine volume | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Uterine volume obtained through ultrasound measurement; The size and shape of the organs are measured by a professional ultrasound physician from our hospital. The volume is calculated using the formula: V=(π /6)*length*anteroposterior diameter*transverse diameter, with the unit being cubic centimeters (cm³).
ovarian volume | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Ovarian volume obtained through ultrasound measurement The size and shape of the organs are measured by a professional ultrasound physician from our hospital. The volume is calculated using the formula: V=(π /6)*length*anteroposterior diameter*transverse diameter, with the unit being cubic centimeters (cm³).
follicle diameter | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Follicle diameter obtained through ultrasound measurement The size and shape of the organs are measured by a professional ultrasound physician from our hospital.
Breast Tanner staging | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Breast Tanner staging (obtained by the physician through physical examination). The Tanner staging criteria and standard illustrations are used for definition. Some obese girls may find it difficult to distinguish between breast tissue and fat tissue, so we have all the subjects raise their arms and have professional doctors use visual and palpation methods to assess the breast development stage.
HbA1c | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Glycated Hemoglobin(detected from the blood). Blood samples are collected from all patients in the morning after an overnight fast. Levels are measured using chemiluminescent immunoassay.
TC | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Total Cholesterol, detected from the blood. Blood samples are collected from all patients in the morning after an overnight fast. Levels are measured using chemiluminescent immunoassay.
TG | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Triglycerides, detected from the blood. Blood samples are collected from all patients in the morning after an overnight fast. Levels are measured using chemiluminescent immunoassay.
LDL-C | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Low-Density Lipoprotein Cholesterol, detected from the blood. Blood samples are collected from all patients in the morning after an overnight fast. Levels are measured using chemiluminescent immunoassay.
HDL-C | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  High-Density Lipoprotein Cholesterol, detected from the blood. Blood samples are collected from all patients in the morning after an overnight fast. Levels are measured using chemiluminescent immunoassay.
ApoB | The measurement times are before the start of the experiment, the 12th week after the start, and the 24th week after the start.
  Apolipoprotein B, detected from the blood. Blood samples are collected from all patients in the morning after an overnight fast. Hormone levels are measured using chemiluminescent immunoassay.

IPD SHARING:
Plan to Share IPD: Undecided